CLINICAL TRIAL: NCT05524558
Title: Assessment of the Hemodynamic Effects of PEEP According to Alveolar Recruitment During the ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Professor, Bicetre Hospital
Other Study IDs: 2022-A00058-35
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: ARDS, Human; Ventilation Therapy; Complications; Alveolar; Disorder
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pulmonary artery catheter — PAC already in place
Device: Esophagal pressure — Esophagal pressure already in place

SUMMARY:
The corner stone of the treatment of ARDS is mechanical ventilation with high levels of positive end-expiratory pressure, also called PEEP. A high level of PEEP is recommended and frequently used. But PEEP can lower cardiac output and contribute to circulatory failure during mechanical ventilation. Nevertheless, in theory, the PEEP-induced pulmonary vascular resistance (PVR) increase could depend on the level of alveolar recruitment, but it has never been proven. Thus, the aim of this study is to determine the relation between the high-PEEP induced PVR and the alveolar recruitment or overdistension.

DETAILED DESCRIPTION:
During acute respiratory distress syndrome (ARDS) the application of positive end-expiratory pressure (PEEP) prevents expiratory alveolar collapse. However, it can induce a predominant recruitment effect or, on the contrary, alveolar overdistension. The recruitment/overdistension ratio can be easily assessed using R/I ratio (or recruitment-to-inflation ratio). However, PEEP is likely to lower cardiac output and contribute to the cardiovascular failure that often occurs in patients with ARDS. Among its hemodynamic effects, PEEP is likely to increase pulmonary vascular resistance and, thus, right ventricular afterload. In theory, this effect should only occur if PEEP over-distends the lung volume, compressing the "extra-alveolar" vessels and increasing their resistance. However, this different effect of PEEP on pulmonary vascular resistance depending on the degree of recruitment or overdistension has never been demonstrated during ARDS in humans.

We retrospectively studied data collected from patients with ARDS, monitored by pulmonary artery catheter (PAC), to eventually find a correlation between the high PEEP-induced PVR increase and recruitement/overdistension profile.

ELIGIBILITY:
Inclusion Criteria:

* ARDS diagnosed
* Invasive mechanical ventilation
* Pulmonary artery catheter already in place
* Esophagal pressure measure

Exclusion Criteria:

* Pregnancy
* Prone position at inclusion
* Legal protection measures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients over the age of 18, exhibiting ARDS and with a PAC-monitoring already in place.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between PVR and recruitment-to-inflation ratio | Up to hospital discharge (maximum : day 60)
  PVR collected at two levels of PEEP and the R/I ratio to assess a relationship between the two variables

SECONDARY OUTCOMES:
Relationship between the R/I ratio and blood gas analysis | Up to hospital discharge (maximum : day 60)
  Data collected from the daily blood samples, to assess a relationship between R/I and arterial oxygen pressure
Relationship between the R/I ratio and respiratory system compliance | Up to hospital discharge (maximum : day 60)
  Ventilatory parameters collected at two levels of PEEP and R/I collected every day to assess a correlation between R/I and lung compliance
Relationship between right ventricle size and R/I ratio | Up to hospital discharge (maximum : day 60)
  Echocardiographic data collected at two levels of PEEP and R/I collected every day to assess a relationship between R/I and changes in RV surface.
Relationship between PVR change and Transpulmonary gradient (TPG) according to R/I | Up to hospital discharge (maximum : day 60)
  Data collected from PAC and R/I measure every day to assess the relationship between R/I and TPG at two levels of PEEP.

CONTACTS AND LOCATIONS:
Locations (1):
- Bicetre Hospital, Le Kremlin-Bicêtre, Île-de-France Region, France

REFERENCES:
- [Background] Michard F, Chemla D, Richard C, Wysocki M, Pinsky MR, Lecarpentier Y, Teboul JL. Clinical use of respiratory changes in arterial pulse pressure to monitor the hemodynamic effects of PEEP. Am J Respir Crit Care Med. 1999 Mar;159(3):935-9. doi: 10.1164/ajrccm.159.3.9805077. PMID 10051276
- [Background] GUYTON AC, LINDSEY AW, ABERNATHY B, RICHARDSON T. Venous return at various right atrial pressures and the normal venous return curve. Am J Physiol. 1957 Jun;189(3):609-15. doi: 10.1152/ajplegacy.1957.189.3.609. No abstract available. PMID 13458395
- [Background] Goldberg HS, Rabson J. Control of cardiac output by systemic vessels. Circulatory adjustments to acute and chronic respiratory failure and the effect of therapeutic interventions. Am J Cardiol. 1981 Mar;47(3):696-702. doi: 10.1016/0002-9149(81)90557-9. No abstract available. PMID 7008571
- [Background] Potkin RT, Hudson LD, Weaver LJ, Trobaugh G. Effect of positive end-expiratory pressure on right and left ventricular function in patients with the adult respiratory distress syndrome. Am Rev Respir Dis. 1987 Feb;135(2):307-11. doi: 10.1164/arrd.1987.135.2.307. PMID 3544983
- [Background] WHITTENBERGER JL, McGREGOR M, BERGLUND E, BORST HG. Influence of state of inflation of the lung on pulmonary vascular resistance. J Appl Physiol. 1960 Sep;15:878-82. doi: 10.1152/jappl.1960.15.5.878. No abstract available. PMID 13784949
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034